CLINICAL TRIAL: NCT02496013
Title: Radiation Dosimetry, Plasma Pharmacokinetics, Biodistribution, Safety and Diagnostic Performance of 68Ga-NEB in Healthy Volunteers and Patients With Hepatic Space-occupying Lesions and Suspicious Lymph Nodes Metastasis
Brief Title: Clinical Translation of a Novel Albumin-Binding PET Radiotracer 68Ga-NEB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM007; ZIAEB000073 (NIH)
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Arteriovenous Malformation; Hemangioma; Neoplasms Lymph Nodes; Lymphedema
MeSH Terms: conditions — Arteriovenous Malformations; Hemangioma; Lymphedema | interventions — 68Ga-1,4,7-triazacyclononane-N,N',N''-triacetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-NEB injection and PET/CT scan (Experimental): Patients for blood pool imaging:
  The patients were intravenously injected with 68Ga-NEB and underwent PET/CT scan 30~45min after the injection.
  Patients for lymph node imaging:
  The patients were locally injected 10~20MBq 68Ga-NEB and followed by dynamic regional PET acquisitions.
  Interventions: Drug: 68Ga-NEB

INTERVENTIONS:
Drug: 68Ga-NEB — 68Ga-NEB were injected into the patients before the PET/CT scans
  Other Names: 68Ga-NOTA conjugated truncated form of Evans blue

SUMMARY:
This is an open-label whole-body PET/CT study for investigation of radiation dosimetry, plasma pharmacokinetics, biodistribution, safety and diagnostic performance of 68Ga-NEB in healthy volunteers and patients with suspected infection. Changes of routine blood and urine tests and any adverse events will be collected from the volunteers. Adverse events will also be observed in the patients.

DETAILED DESCRIPTION:
The labeling of albumin has advantages as drawing blood is unnecessary and the operator labeling is not exposed to potentially infectious material. Evans blue (EB) dye has high affinity for serum albumin, The final obtained products NEB (a NOTA conjugate of a truncated form of Evans blue for in vivo albumin labeling) was proceeded strict quality controls.

No fasting, hydration or other specific preparation was requested on the day of imaging.

Patients for blood pool imaging underwent whole-body PET/CT acquisitions 30-45 min after intravenous injection of 111-148 MBq (3-4 mCi) 68Ga-NEB with each bed position lasted for 2 min and a standard routine 18F-FDG PET/CT within one week.

Patients for lymph node imaging including the breast nodules patients underwent a standard routine 18F-FDG PET/CT first, and were locally injected 10~20MBq 68Ga-NEB, followed by dynamic chest regional PET acquisitions.

A Siemens MMWP workstation was used for post-processing. Visual analysis was used to determine the general biodistribution and the temporal and intersubject stability. Semiquantitative methods were applied for image analysis.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide a written informed consent
* Males and females, ≥18 years old；
* Diagnostic CT or MRI suggesting a diagnosis of liver focal lesion(s). In suspicion of arteriovenous malformations. Newly diagnosed breast cancer and lymph node metastasis is not clear. The tumor will be surgically removed and histological diagnosis will be available. Evaluation of cardiac function.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential；
* Known severe allergy or hypersensitivity to IV radiographic contrast；
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the investigator, may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of 68Ga-NEB as determined by standardized uptake value for PET imaging | 1 years

SECONDARY OUTCOMES:
Adverse events collection | 2 week
  Adverse events within 2 weeks after the injection and scanning of healthy volunteers and patients will be followed and assessed
Routine blood test | 24 hours
  Routine blood test of healthy volunteers will be measured before injection and 24 hours after test
Serum albumin | 24 hours
  Serum albumin of healthy volunteers will be measured before injection and 24 hours after test
Routine urine test | 24 hours
  Routine urine test of healthy volunteers will be measured before injection and 24 hours after test
Assessment of liver lesions as determined by standardized uptake value of 68Ga-NEB PET | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, Dr., Study Chair — Peking Union Medical College Hospital
Locations (1):
- PET centre, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No